CLINICAL TRIAL: NCT00995527
Title: Characterization of the Innate Immune Response in Healthy NIH Employees at Baseline and After Immunization With the H1N1 Vaccine
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090245; 09-H-0245
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-06-25

CONDITIONS: Healthy Volunteers
Keywords: Post Swine Flu Blood Samples; Biologic Sample Collection; Laboratory Research Samples; H1N1 Vaccine Samples; HV; Healthy Volunteer

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The Center for Human Immunology, Autoimmunity, and Inflammatory Diseases is conducting research investigating how the swine flu (H1N1) vaccine affects the immune system. The exposure to the new swine flu vaccine gives us a rare opportunity to learn about how the human immune system responds to a new vaccine.
* Researchers are interested in collecting blood samples from individuals who have received the vaccine. Participants will be selected from a group of healthy volunteers who will be receiving the H1N1 vaccine because it is mandatory for their work at the National Institutes of Health. This protocol will be one of the first studies to characterize the human innate immune response to H1N1 vaccine.

Objectives:

- To collect blood samples for research purposes before and after participants receive a standard non-research vaccination against swine flu (H1N1).

Eligibility:

* Healthy individuals 18 years of age and older who are employees of the National Institutes of Health.
* Individuals who have had confirmed cases of influenza in the past year are not eligible to participate.

Design:

* Participants will be admitted for a 36-hour inpatient stay, during which blood samples will be taken frequently. Participants will have a standard intravenous catheter (similar to the one used for intravenous infusions) put in place to avoid multiple needle sticks.
* Participants will be assigned into one of two groups; the two groups differ in the timing of blood draws but not in the overall amount of blood drawn.
* Group 1: Blood samples 30 minutes before and immediately before vaccination. Additional samples will be taken 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 30, and 36 hours after vaccination.
* Group 2: Blood samples 30 minutes before and immediately before vaccination. Additional samples will be taken over the following 36 hours, with exact timing to be determined based on the findings from group 1.
* All participants will provide blood samples 7 days after being released from the inpatient stay.
* Because of the amount of blood being drawn for research, participants should not donate blood or take part in any other protocols that collect blood while participating in this study.

DETAILED DESCRIPTION:
Seasonal influenza is a major health problem whose impact is typically reduced by vaccination. The H1N1 (swine flu) influenza virus is an emerging pathogen which has the potential to cause devastating morbidity and mortality in the coming months. In June 2009, the World Health Organization declared the H1N1 outbreak to be a global pandemic. At present there are limited data on the early non-specific (innate) immune responses in adult recipients of the H1N1 vaccine.

Therefore the Center for Human Immunology, Autoimmunity, and Inflammatory Diseases proposes this protocol designed to investigate the early innate immune response. Healthy adult subjects (NIH employees) will be admitted as inpatients to receive the FDA-licensed H1N1 vaccine followed by serial blood draws. These samples will be used to perform comprehensive and detailed analyses of the innate immune system s response to vaccination. To our knowledge, this protocol will be the first study to characterize the human innate immune response to H1N1 vaccine. This information may be useful in designing newer, more effective vaccines to prevent the spread of H1N1.

The primary objective is to collect blood to be used strictly for laboratory studies designed to characterize the innate immune response to H1N1 vaccine. Samples will be collected from healthy adult volunteers (NIH employees) at baseline and serially during the first 36 hours after vaccination with the H1N1 vaccine.

ELIGIBILITY:
* INCLUSION CRITERIA:
* NIH employees scheduled to receive the H1N1 vaccine through OMS
* Healthy status confirmed by History, Physical Exam and blood work through the CHI Screening Protocol
* Age 18 years and older (no upper limit)
* Able to comprehend the investigational nature of the protocol and provide informed consent

EXCLUSION CRITERIA:

* Recipient of another vaccine or immune modulating drug within 6 months prior to study entry. Seasonal influenza vaccine may be administered up to 3 days prior to enrollment or after completion of study participation (day 7 blood draw)
* Confirmed influenza within the past 1 year
* Severe allergies to eggs or their products
* Prior severe reactions to vaccines
* Participation on any blood collection or blood donation procedure during study that will bring the total blood draw > 550m1 over 8 weeks.
* Current pregnancy (women of child bearing potential must have a negative serum pregnancy test done on screening within 1 week of protocol accrual)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09-30; Study Completion 2014-06-25

PRIMARY OUTCOMES:
Results of research laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Shira Y Perl, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Neumann G, Noda T, Kawaoka Y. Emergence and pandemic potential of swine-origin H1N1 influenza virus. Nature. 2009 Jun 18;459(7249):931-9. doi: 10.1038/nature08157. PMID 19525932
- [Background] Zimmer SM, Burke DS. Historical perspective--Emergence of influenza A (H1N1) viruses. N Engl J Med. 2009 Jul 16;361(3):279-85. doi: 10.1056/NEJMra0904322. Epub 2009 Jun 29. No abstract available. PMID 19564632